CLINICAL TRIAL: NCT02517918
Title: Metronomic Cyclophosphamide and Methotrexate Combined With Zoledronic Acid and Sirolimus in Patients With Advanced Solid Tumor With Bone Metastasis and Advanced Pretreated Osteosarcoma. A Phase Ib Study From the French Sarcoma Group
Brief Title: Metronomic Chemotherapy in Patients With Advanced Solid Tumor With Bone Metastasis and Advanced Pretreated Osteosarcoma
Acronym: METZOLIMOS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Reliable Cancer Therapies (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IB 2014-01
Record Dates: First submitted 2015-02-19; First posted 2015-08-07 (Estimated); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor; Osteosarcoma
Keywords: Advanced solid tumor; Bone metastasis and advanced pretreated osteosarcoma; Phase I trial; Dose escalation and expansion cohort; Biomarkers study
MeSH Terms: conditions — Osteosarcoma | interventions — Cyclophosphamide; Methotrexate; Sirolimus; Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: This is a prospective open-labeled phase I trial based on :
  * a dose escalating study design assessing two dose levels of sirolimus when prescribed in combination with metronomic cyclophosphamide (CP), methotrexate (MT) and zoledronic acid (ZA)
  * an expansion cohort once the MTD is established.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus combined with CP, MT and ZA (Experimental): Drug : Metronomic Cyclophosphamide, Methotrexate, Sirolimus, Zoledronic acid Assessment of the maximum tolerated dose of sirolimus Cyclophosphamide, Methotrexate and Sirolimus will be administrated orally. Zoledronic Acid will be administrated by infusion (IV).
  Interventions: Drug: Sirolimus combined with CP, MT and ZA

INTERVENTIONS:
Drug: Sirolimus combined with CP, MT and ZA — Cyclophosphamide, Methotrexate and Sirolimus will be administrated orally. Zoledronic Acid will be administrated by infusion (IV).
  Trial based on a dose escalating study design assessing two dose levels of sirolimus when prescribed in combination with metronomic cyclophosphamide (CP), methotrexate (MT) and zoledronic acid (ZA) followed by an expansion cohort once the MTD is established.
  Other Names: Endoxan, Methotrexate, Rapamune, Zoledronic acid

SUMMARY:
This is a prospective open-labeled phase I trial based on a dose escalating study design assessing two dose levels of sirolimus when prescribed in combination with metronomic cyclophosphamide (CP), methotrexate (MT) and zoledronic acid (ZA) followed by an expansion cohort once the Maximum Tolerated Dose (MTD) is established.

DETAILED DESCRIPTION:
The dose escalation part of the trial will be concerned on adults with advanced solid tumor with bone metastasis and young and adult patients with unresectable locally advanced or metastatic osteosarcoma.

The Expansion cohort will be conducted on young and adult patients with unresectable locally advanced or metastatic osteosarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histology:

   * Advanced solid tumor with radiologically proven bone metastasis, (dose escalation part)
   * Patients with osteogenic osteosarcoma (dose escalation part and expansion cohort) histologically confirmed by central review
2. Metastatic or unresectable locally advanced disease, not eligible for alternative local treatment (radiotherapy for instance)
3. Age > 18 years for patients with solid tumor and ≥ 13 years for patients with osteosarcoma
4. ECOG, performance status ≤ 1
5. Life expectancy > 3 months
6. Measurable disease according to RECIST v1.1. At least one site of disease must be uni-dimensionally ≥ 10 mm
7. Patients must have histologically confirmed diagnosis of locally advanced and/or metastatic solid tumors, which are not amenable to standard treatment, including for patients with osteosarcoma conventional agents such as anthracyclines, platinum salts, ifosfamide and/or methotrexate
8. At least three weeks since last chemotherapy, immunotherapy or any other pharmacological treatment and/or radiotherapy
9. Adequate haematological, renal, metabolic and hepatic function:

   * Haemoglobin ≥ 10 g/dl (patients may have received prior red blood cell transfusion, if clinically indicated); leucocytes ≥ 3 x 10^9/l, absolute neutrophil count ≥ 1.5 x 10^9/l, and platelet count ≥ 120 x 10^9/l.
   * Alanine aminotransferase and aspartate aminotransferase ≤ 2.5 x upper limit of normality (ULN)
   * Total bilirubin ≤ 1.5 x ULN
   * Calculated creatinine clearance > 40 ml/min/1.73 m² (according to MDRD formula)
   * Creatine phosphokinase ≤ 2.5 x ULN
   * Albumin > 25 g/l
10. No prior or concurrent malignant disease diagnosed or treated in the last 2 years except adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma,
11. Recovery to grade ≤ 1 from any adverse event derived from previous treatment (excluding alopecia of any grade and non-painful peripheral neuropathy grade ≤ 2) according to the NCI-CTCAE, version 4
12. Patients with a French social security in compliance with the French law relating to biomedical research
13. Voluntarily signed and dated written informed consent prior to any study specific procedure
14. Women of childbearing potential must have a negative serum pregnancy test before study entry. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for six months after discontinuation of treatment

Exclusion Criteria:

1. Previous treatment with sirolimus
2. Concomitant diseases/conditions:

   * Clinically significant and/or rapidly accumulating ascites, pericardial and/or pleural effusions
   * Unstable cardiac disease, pulse oximetry saturation < 90% at rest
   * Clinically significant immunodeficiency, such as HIV or active Hepatitis B or C
   * History of auto-immune disease, transplantation
3. Central nervous system malignancy
4. Men or women of childbearing potential who are not using an effective method of contraception; women who are pregnant or breast feeding
5. Patients receiving any substances that are inhibitors or inducers of CYP450 3A4
6. Ongoing or recent (<6 weeks) dental problem, including any severe tooth or jaw infection (mandible and maxilla), dental trauma, dental or stomatological surgery (implants). Current dental cares are allowed
7. History of maxillary osteonecrosis or delayed healing after dental surgery
8. Participation to a study involving a medical or therapeutic intervention in the last 30 days
9. Previous enrolment in the present study
10. Patient unable to follow and comply with the study procedures because of any geographical, familial, social or psychological reasons
11. Known hypersensitivity to any involved study drug or any of its formulation components
12. Patients receiving live vaccines within 30 days prior to the first dose of study therapy and while participating in study

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-09-05 (Actual); Study Completion 2021-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maud TOULMONDE, Doctor, Study Chair — Institut Bergonié
Locations (3):
- France (3):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: February 16th, 2015 and last patient enrolled: March 11th, 2021
Groups:
- Dose Escalation Part With Sirolimus (Si) Dose 4 mg: Prospective open-labeled phase I trial. The dose escalation design to identify the maximum tolerated dose will be the traditional 3+3 design.
  Sirolimus (SI) dose 4 mg when prescribed in combination with metronomic cyclophosphamide (CP), methotrexate (MT) and zoledronic acid (ZA) Sirolimus will be administered per os once daily, continuously. One cycle consits of 28 days.
  Number of subjects : 6. Cyclophosphamide will be administered per os bi-daily (50 mg x 2), and given on a week on/week off schedule.
  Methotrexate will be administered per os bi-daily (2.5 mg x 2), and given on day 1 and 4 every week.
  Zoledronic acid will be administered at home by intravenous infusion (4 mg) on Day 2 of each cycle, every 4 weeks.
- Dose Escalation Part With Sirolimus (SI) Dose 6 mg: Prospective open-labeled phase I trial. The dose escalation design to identify the maximum tolerated dose will be the traditional 3+3 design.
  Sirolimus (SI) dose 6 mg when prescribed in combination with metronomic cyclophosphamide (CP), methotrexate (MT) and zoledronic acid (ZA) Sirolimus will be administered per os once daily, continuously. One cycle consits of 28 days.
  Number of subjects : 3. Cyclophosphamide will be administered per os bi-daily (50 mg x 2), and given on a week on/week off schedule.
  Methotrexate will be administered per os bi-daily (2.5 mg x 2), and given on day 1 and 4 every week.
  Zoledronic acid will be administered at home by intravenous infusion (4 mg) on Day 2 of each cycle, every 4 weeks.
- Expansion Cohort With Dose Sirolimus (SI) 4 mg: Prospective open-labeled phase I trial. The expansion cohort is designed to enable to detect antitumor activity observed with sirolimus (SI) combined with cyclophosphamide (CP), methotrexate (MT) and zoledronic acid (ZA).
  Sirolimus (SI) dose 4 mg when prescribed in combination with metronomic cyclophosphamide (CP), methotrexate (MT) and zoledronic acid (ZA) Sirolimus will be administered per os once daily, continuously. One cycle consits of 28 days.
  Number of subjects : 14. Cyclophosphamide will be administered per os bi-daily (50 mg x 2), and given on a week on/week off schedule.
  Methotrexate will be administered per os bi-daily (2.5 mg x 2), and given on day 1 and 4 every week.
  Zoledronic acid will be administered at home by intravenous infusion (4 mg) on Day 2 of each cycle, every 4 weeks.
Period: Overall Study
Arm/Group | Dose Escalation Part With Sirolimus (Si) Dose 4 mg | Dose Escalation Part With Sirolimus (SI) Dose 6 mg | Expansion Cohort With Dose Sirolimus (SI) 4 mg
Started | 6 | 3 | 14
Completed (Population assessable : Dose escalation part (tolerance) : Patients who received at least one dose of one of the trial's products and have received the complete C1 cycle (28 days: D1 to D28) or have exhibited a DLT during C1. Expansion cohort (efficacy) : Patients eligible and who received at least one complete or two incomplete treatment cycles and least one disease measurement recorded not less than eight weeks after treatment onset.) | 6 | 3 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients included, regardless of whether or not treatment was administered, and regardless violations of any eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Part With Sirolimus (Si) Dose 4 mg | Dose Escalation Part With Sirolimus (SI) Dose 6 mg | Expansion Cohort With Dose Sirolimus (SI) 4 mg | Total
Number analyzed (Participants) | 6 | 3 | 14 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (13.1) | 65.4 (12) | 36.3 (21.4) | 44.3 (21.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6 | 12
  Male | 2 | 1 | 8 | 11
Region of Enrollment [Number; unit: participants]
  France | 6 | 3 | 14 | 23

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Part: Number of Dose-Limiting Toxicities (DLTs) at Each Dose Level on Cycle 1
Description: A DLT is defined as an adverse event (AE) or laboratory abnormality that fulfills the criteria below:
  * Is considered to be at least possibly related to the study treatment
  * Occurs during the first cycle of treatment
  * Is unrelated to disease, disease progression, inter-current illness, or concomitant medications
  * Meets one of the criteria below, graded as outlined or according to NCI CTCAEv4.3:
    * Grade 4 non-haematological toxicity (not laboratory)
    * Grade 3 non-haematological toxicity > 3 days (not laboratory) (except for asthenia, 1rst episode of nausea/vomiting without maximal symptomatic/prophylactic treatment)
    * Grade ≥ 3 non-hematologic laboratory value if medical intervention is required to treat the patient, or the abnormality leads to hospitalization, or the abnormality persists for > 1 week
    * Grade ≥ 3 hematologic toxicity > 3 days (except for lymphopenia)
    * Grade 4 lymphopenia
    * Confirmed febrile neutropenia
Time Frame: During the first cycle (28 days)
Population: Population assessable : Patients who received at least one dose of one of the trial's products and have received the complete C1 cycle (28 days: D1 to D28) or have exhibited a DLT during C1.
Measure: Number; unit: Number of DLTs
Arm/Group | Dose Escalation Part With Sirolimus (Si) Dose 4 mg | Dose Escalation Part With Sirolimus (SI) Dose 6 mg
Number analyzed (Participants) | 6 | 3
Number of DLTs | 0 | 2

2. Primary Outcome: Expansion Cohort : Antitumor Activity Observed With Sirolimus Combined With CP, MT and ZA, in Terms of 6-month Non-progression Rate
Description: 6-month non-progression rate defined as the rate of complete or partial response or stable disease at 6 months using RECIST v1.1 :
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions and also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD
  * Unevaluable : patients stopped the treatment before tumor assessment.
Time Frame: 6-month non-progression rate as per RECIST v1.1
Population: Population assessable : Patients eligible and who received at least one complete or two incomplete treatment cycles and least one disease measurement recorded not less than eight weeks after treatment onset.
Measure: Number; unit: participants
Arm/Group | Expansion Cohort With Dose Sirolimus (SI) 4 mg
Number analyzed (Participants) | 14
participants
  Complete response | 0
  Partial response confirmed | 1
  Stable disease | 1
  Progression | 10
  Unevaluable according to RECIST v1.1 | 2

3. Secondary Outcome: Dose Escalation Part : Antitumor Activity Observed With Sirolimus Combined With CP, MT and ZA, Best Objective Response Rate (ORR) as Per RECIST v1.1
Description: The best objective response (BOR) is the best response recorded for each patient from the start of the study treatment until the end of treatment for progressive disease, death, patient or investigator decision.
  BOR is determined by investigator review of tumor assessments using RECIST v1.1 :
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions and also demonstrate an absolute increase of at least 5 mm
  * Stable Disease (SD)
  Tumor assessment were repeated every 8 weeks (±7 days, i.e Week 8, 16, 24, etc.) from start of treatment and at least 4 weeks after the first CR or PR, even if there are treatment delays, average of 4 months
Time Frame: Tumor assessment were repeated every 8 weeks (±7 days, i.e Week 8, 16, 24, etc.) from the start of treatment and at least 4 weeks after the first CR or PR, even if there are treatment delays, an average of 4 months.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Dose Escalation Part With Sirolimus (Si) Dose 4 mg | Dose Escalation Part With Sirolimus (SI) Dose 6 mg
Number analyzed (Participants) | 6 | 3
participants
  Completed response | 0 | 0
  Partial response | 0 | 0
  Stable disease | 3 | 1
  Progression | 2 | 1
  Inevaluable for response | 1 | 1

4. Secondary Outcome: Dose Escalation Part : Antitumor Activity Observed With Sirolimus Combined With CP, MT and ZA, 1-year Progression-free Survival (PFS)
Description: 1-year Progression-free survival (PFS) is defined as the time from study treatment initiation to the first occurrence of disease progression, as determined by investigator review of tumor assessments using RECIST v1.1, or death from any cause during the study (i.e., within 30 days after the last dose of study treatment).
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: 1-year Progression-free survival (PFS) as per RECIST v1.1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part With Sirolimus (Si) Dose 4 mg | Dose Escalation Part With Sirolimus (SI) Dose 6 mg
Number analyzed (Participants) | 6 | 3
Participants | 6 | 1

5. Secondary Outcome: Dose Escalation Part : Antitumor Activity Observed With Sirolimus Combined With CP, MT and ZA, 1-year Overall Survival (OS)
Description: 1-year Overall Survival (OS) is defined as the time from first infusion to death (of any cause)
Time Frame: 1-year Overall Survival (OS) as per RECIST v1.1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part With Sirolimus (Si) Dose 4 mg | Dose Escalation Part With Sirolimus (SI) Dose 6 mg
Number analyzed (Participants) | 6 | 3
Participants | 3 | 0

6. Secondary Outcome: Expansion Cohort : Antitumor Activity Observed With Sirolimus Combined With CP, MT and ZA, Best Objective Response Rate (ORR) as Per RECIST v1.1
Description: The best objective response (BOR) is the best response recorded for each patient from the start of the study treatment until the end of treatment for progressive disease, death, patient or investigator decision.
  BOR is determined by investigator review of tumor assessments using RECIST v1.1 :
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions and also demonstrate an absolute increase of at least 5 mm
  * Stable Disease (SD) Tumor assessment were repeated every 8 weeks (±7 days, i.e Week 8, 16, 24, etc.) from start of treatment and at least 4 weeks after the first CR or PR, even if there are treatment delays, an average of 4 months
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Expansion Cohort With Dose Sirolimus (SI) 4 mg
Number analyzed (Participants) | 14
participants
  Complete response | 0
  Confirmed Partial response | 1
  Stable disease | 3
  Progression | 8
  Inevaluable for response | 2

7. Secondary Outcome: Expansion Cohort : Antitumor Activity Observed With Sirolimus Combined With CP, MT and ZA, 1-year Progression-free Survival (PFS) as Per RECIST v1.1
Description: as for outcome 4
Time Frame: 1-year Progression-free survival (PFS) as per RECIST v1.1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Expansion Cohort With Dose Sirolimus (SI) 4 mg
Number analyzed (Participants) | 14
months | 1.8 [1.4 to 3.6]

8. Secondary Outcome: Expansion Cohort : Antitumor Activity Observed With Sirolimus Combined With CP, MT and ZA, 1-year Overall Survival (OS) as Per RECIST v1.1
Description: 1-year Overall Survival (OS) is defined as the time from first infusion to death (of any cause)
Time Frame: 1-year Overall Survival (OS) as per RECIST v1.1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort With Dose Sirolimus (SI) 4 mg
Number analyzed (Participants) | 14
Participants | 7

ADVERSE EVENTS:
Time Frame: Safety profile was continuously followed : monitored every 28 days during treatment consultation and up to 30 days after the last treatment administration or until the start of a new antitumor therapy, whichever occurs first. In case of SAE, monitoring could be improved as per investigator's judgement. After treatment discontinuation, patients were followed up 4 weeks later for toxicities. Grade 3 or 4 toxicity were monitored until resolution, through study completion, an average of 13 months.
Description: Safety population: all patients having received at least one treatment administration.
  All adverse events (related and unrelated to treatment) are reported. All serious adverse events (related and unrelated to treatment) are reported.
  Adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE).
Arm/Group | Dose Escalation Part With Sirolimus (Si) Dose 4 mg | Dose Escalation Part With Sirolimus (SI) Dose 6 mg | Expansion Cohort With Dose Sirolimus (SI) 4 mg
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/3 | 9/14
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Part With Sirolimus (Si) Dose 4 mg (N=6) | Dose Escalation Part With Sirolimus (SI) Dose 6 mg (N=3) | Expansion Cohort With Dose Sirolimus (SI) 4 mg (N=14)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Musculoskeletal chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (7) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 2 (2) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 3 (5)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Part With Sirolimus (Si) Dose 4 mg (N=6) | Dose Escalation Part With Sirolimus (SI) Dose 6 mg (N=3) | Expansion Cohort With Dose Sirolimus (SI) 4 mg (N=14)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 4 (6)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (5) | 2 (2) | 6 (8)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 3 (3) | 6 (6)
Fever (General disorders) | 1 (1) | 0 (0) | 4 (4)
Flu like symptoms (General disorders) | 2 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Gum infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 5 (5)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 2 (2) | 4 (4)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 1 (1) | 0 (0) | 0 (0)
GGT increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2) | 1 (1) | 6 (6)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (3) | 2 (2)
Platelet count decreased (Investigations) | 2 (2) | 3 (3) | 7 (8)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
WORSENING OF GENERAL STATUS (General disorders) | 1 (1) | 0 (0) | 0 (0) — General disorders and administration site conditions - Other, specify
INFLAMMATORY SYNDROM (General disorders) | 0 (0) | 0 (0) | 2 (2) — General disorders and administration site conditions - Other, specify
HOT FLUSHES (General disorders) | 0 (0) | 0 (0) | 1 (1) — General disorders and administration site conditions - Other, specify
POLYDYPSIA (General disorders) | 0 (0) | 0 (0) | 1 (1) — General disorders and administration site conditions - Other, specify
ALTERATION OF GENERAL STATUS (General disorders) | 0 (0) | 0 (0) | 1 (1) — General disorders and administration site conditions - Other, specify
LDH INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) — Investigations - Other, specify
CRP INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) — Investigations - Other, specify
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — Metabolism and nutrition disorders - Other, specify
SUBCUTANEOUS NODULE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) — Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify
DYSURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Renal and urinary disorders - Other, specify
NOCTURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Renal and urinary disorders - Other, specify
URINARY DISORDERS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Renal and urinary disorders - Other, specify
POLYURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Renal and urinary disorders - Other, specify
VAGINAL ULCERATION (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — Reproductive system and breast disorders - Other, specify
ESCHAR OF THE SACRUM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Skin and subcutaneous tissue disorders - Other, specify

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT02517918/SAP_000.pdf